CLINICAL TRIAL: NCT05900245
Title: To Explore the Influence of Different Anesthesia Induction Schemes on the Quality and Clinical Effect of Electroconvulsive Convulsions in Patients With Depression Based on EEG Monitoring
Brief Title: Anesthesia Induction Schemes of Electroconvulsive Convulsions in Patients With Depression Based on EEG Monitoring
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Min Su (Other)
Responsible Party: Sponsor-Investigator, Min Su, Professor of Anesthesiology, First Affiliated Hospital of Chongqing Medical University
Organization: First Affiliated Hospital of Chongqing Medical University (Other)
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Supportive Care
Other Study IDs: CQMUFH-2023-052
Record Dates: First submitted 2023-03-09; First posted 2023-06-12 (Actual); Last update posted 2024-01-26 (Actual); Status verified 2024-01

CONDITIONS: Depression; Electroconvulsive Therapy; Electroencephalography
Keywords: Depression,Electroconvulsive Therapy,Electroencephalography
MeSH Terms: conditions — Depression

STUDY DESIGN:
Intervention Model Description: Due to the fact that anesthesiologists need to determine the timing of electrical stimulation based on the level of consciousness index during the treatment of electric shock, this study is a randomized controlled, single blind study.Due to the varying frequency of electroconvulsive therapy performed by each subject, with an average of 6-12 times and varying duration of each electroconvulsive treatment, this study uses a mixed effects model to analyze the relationship between different consciousness indices and patient factors on the duration of EEG seizures.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Due to the fact that anesthesiologists need to determine the timing of electrical stimulation based on the level of consciousness index during the treatment of electric shock, this study is a randomized controlled, single blind study. The subjects were not aware of their grouping, consciousness index level, and the anesthesiologist was aware of the subjects' consciousness index level, but did not participate in data analysis. The data analyst is not clear about the specific content of the grouping.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group H：IoC1 60-70 (Active Comparator): This study used an EEG bispectral index monitor (Apolo 9000A) to monitor consciousness index 1 (IoC1) and consciousness index 2 (IoC2) before electric shock, and then induced anesthesia with propofol 1.5mg/kg and succinylcholine 1mg/kg， following by mask pressurized oxygen supply，dental pads protect the tongue and monitoring the concentration of end-expiratory carbon dioxide. Electrical stimulation is performed when the consciousness index 1 is between 60 and 70. The electrode is located on the bilateral temporal side;Electric shock equipment:ThymatronSystem Ⅳ Electroconvulsive System，manufacturer：SOMATICS, USA；Propofol manufacturer: AstraZeneca of the UK, concentration: 10mg/ml. Succinylcholine manufacturer: Shanghai Xudong Haipu Pharmaceutical Co., Ltd.China, concentration: 2ml: 0.1g.
  Interventions: Other: Index of consciousness+Anesthetic（propofol）+Muscle relaxant（Succinylcholine）
- Group M: IoC1 50-60 (Active Comparator): This study used an EEG bispectral index monitor (Apolo 9000A) to monitor consciousness index 1 (IoC1) and consciousness index 2 (IoC2) before electric shock, and then induced anesthesia with propofol 1.5mg/kg and succinylcholine 1mg/kg， following by mask pressurized oxygen supply，dental pads protect the tongue and monitoring the concentration of end-expiratory carbon dioxide. Electrical stimulation is performed when the consciousness index 1 is between 50 and 60. The electrode is located on the bilateral temporal side;Electric shock equipment:ThymatronSystem Ⅳ Electroconvulsive System，manufacturer：SOMATICS, USA；Propofol manufacturer: AstraZeneca of the UK, concentration: 10mg/ml. Succinylcholine manufacturer: Shanghai Xudong Haipu Pharmaceutical Co., Ltd.China, concentration: 2ml: 0.1g.
  Interventions: Other: Index of consciousness+Anesthetic（propofol）+Muscle relaxant（Succinylcholine）
- Group L：IoC1 40-50 (Active Comparator): This study used an EEG bispectral index monitor (Apolo 9000A) to monitor consciousness index 1 (IoC1) and consciousness index 2 (IoC2) before electric shock, and then induced anesthesia with propofol 1.5mg/kg and succinylcholine 1mg/kg， following by mask pressurized oxygen supply，dental pads protect the tongue and monitoring the concentration of end-expiratory carbon dioxide. Electrical stimulation is performed when the consciousness index 1 is between 40 and 50. The electrode is located on the bilateral temporal side;Electric shock equipment:ThymatronSystem Ⅳ Electroconvulsive System，manufacturer：SOMATICS, USA；Propofol manufacturer: AstraZeneca of the UK, concentration: 10mg/ml. Succinylcholine manufacturer: Shanghai Xudong Haipu Pharmaceutical Co., Ltd.China, concentration: 2ml: 0.1g.
  Interventions: Other: Index of consciousness+Anesthetic（propofol）+Muscle relaxant（Succinylcholine）

INTERVENTIONS:
Other: Index of consciousness+Anesthetic（propofol）+Muscle relaxant（Succinylcholine） — EEG monitoring is performed before induction of electrical shock anesthesia（propofol1.5mg/kg+Succinylcholine1mg/kg）, and the timing of electrical stimulation is determined based on the level of consciousness index 1 displayed on the EEG.

SUMMARY:
Depression is a common clinical mental disease with high incidence rate, high recurrence rate, high suicide rate and high disability rate. As a first-line treatment for depression with refractory, high suicide risk and obvious psychotic symptoms, electric shock has a definite effect on depression, but may lead to cognitive impairment. The induction of extensive epileptiform discharges in the cerebral cortex by electric shock therapy is the key to ensure the treatment effect. The level of epileptiform discharges in the brain is mainly reflected in the quality of convulsions. The quality of electroconvulsive convulsions is affected by factors such as age, stimulation power, anesthetic drugs and depth of anesthesia. Most anesthetics have anticonvulsive properties, such as barbiturate or propofol, which may have a negative impact on the quality of convulsions, thus affecting the therapeutic effect. If the parameters of electric shock, such as stimulation dose, are modified, although the quality and treatment effect of convulsions can be improved, it may also lead to higher cognitive side effects. The depth of anesthesia also affects the quality and efficacy of electric shock convulsions, and the quality of convulsions is higher when stimulated at a shallow level of anesthesia. However, if the use of narcotic drugs is reduced to improve the quality of convulsions, the risk of restlessness and delirium after electric shock may be higher and the comfort of patients may be lower. Therefore, this study compared the effects of different anesthesia induction schemes on the quality and clinical efficacy of electroconvulsive seizures in patients with depression based on EEG monitoring, and explored the optimal depth of anesthesia.

DETAILED DESCRIPTION:
This study is a randomized controlled, single blind clinical trial comparing the quality of convulsions and clinical effects of electroconvulsive therapy under different levels of consciousness index (IoC).A total of 24 participants were included in this study, all from the inpatient department of the Psychiatric Department of the First Affiliated Hospital of Chongqing Medical University. They were diagnosed as depression patients according to the International Classification of Diseases (ICD-11), and their depression level and cognitive function level were evaluated by trained psychiatrists; In the study, the subjects use the EEG bispectral index monitor (Apollo-9000A) to monitor IoC1(Index of consciousness 1) and IoC2(Index of consciousness 2) before electric shock.Then anesthesia induction was performed using propofol 1.5mg/kg and scoline 1mg/kg. According to the difference in consciousness index 1 (IoC1), the subjects were randomly divided into three groups, namely H group (IoC1 60-70), M group (IoC1 50-60), and L group (IoC1 40-50). All subjects underwent assisted breathing after anesthesia induction, monitoring the concentration of end-expiratory carbon dioxide, and conducting electrical stimulation when the consciousness index reached the corresponding level,and the electrode position is bilateral temporal area. The main outcome measure is EEG seizure duration ,and the secondary outcome measures include average Seizure Energy Index(SEI), electric shock stimulation energy, post-seizure inhibition index, the fastest heart rate, Hamilton Depression Scale (HAMD-24) score, Montreal Cognitive Assessment Scale (MoCA) score, adverse reactions during awakening and the interval between anesthesia induction and the start of electrical stimulation.

Due to the varying frequency of electroconvulsive therapy performed by each subject, with an average of 6-12 times and varying duration of each electroconvulsive treatment, this study uses a mixed effects model to analyze the relationship between different consciousness indices and patient factors on the duration of EEG seizures. The depression score and cognitive function score before and after the complete course of electric shock are compared between groups using LSD-t test.

ELIGIBILITY:
Inclusion Criteria:

* In-patients who meet the diagnostic criteria of moderate and severe depression in the 11th edition of the International Classification of Diseases (ICD-11)
* Age 18-60 years old, gender unlimited
* Primary school or above education level
* Indications for MECT treatment
* Normal hearing and vision (including color discrimination)
* The patient voluntarily participated in the study and signed the informed consent form, and the guardian also signed the informed consent form.

Exclusion Criteria:

* History of physical disease, brain organic disease and abuse of alcohol and psychoactive substances
* Patients with bipolar disorder
* Primary insomnia
* Combined with other mental diseases
* Combined with obesity, diabetes and other metabolic diseases
* Combined with hypertension, cardiovascular disease or cerebrovascular disease
* Combined with Alzheimer's disease
* Pregnant and lactating women.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-06-12 (Actual); Primary Completion 2024-03-31 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
EEG seizure duration | up to 30 minutes after each electroconvulsive treatment
  Duration of EEG convulsions, in seconds,the most important index of the quality of EEG during the treatment of electric shock

SECONDARY OUTCOMES:
average Seizure Energy Index(SEI) | up to 30 minutes after each electroconvulsive treatment
  Indicator of quality of convulsive, in uV2
electric shock stimulation energy | up to 30 minutes after each electroconvulsive treatment
  Indicator of electric shock stimulation energy, in mC
post-seizure inhibition index | up to 30 minutes after each electroconvulsive treatment
  Indicator of quality of convulsive, in %
Bispectral EEG monitoring index | up to 30 minutes after each electroconvulsive treatment
  Depth of sedation and injury stress index,Value range 0-100
Maximun heart rate | up to 30 minutes after each electroconvulsive treatment
  Maximum heart rate during electrical stimulation,in times/minute
Hamilton score | through study completion, an average of 1 year
  Depression score,A total score of 81 points, ≤ 8 points without depression, 8-20 points with possible depression, 20-35 points with mild to moderate depression, ≥ 35 points with severe depression
Montreal cognitive score | through study completion, an average of 1 year
  cognitive function assessment,A total score of 30 points,<26 points determines the presence of cognitive impairment
Recovery period restlessness | up to 4 hours after each electroconvulsive treatment
  Complications during anesthesia recovery，Using Richmond restless sedation scale
Recovery period delirium | up to 4 hours after each electroconvulsive treatment
  Complications during anesthesia recovery，Using CAM-ICU scale
Recovery period nausea and vomiting | up to 4 hours after each electroconvulsive treatment
  Complications during anesthesia recovery，Using index of nausea and vomiting and retching（R-INVR）
Recovery period muscle soreness, headache, dizziness | up to 4 hours after each electroconvulsive treatment
  Complications during anesthesia recovery，Using 0 for none, 1 for yes
interval between anesthesia induction and the start of electrical stimulation | up to 4 hours after each electroconvulsive treatment
  Time to wait for electrical stimulation after administration，in seconds
intraoperative awareness | up to 4 hours after each electroconvulsive treatment
  During general anesthesia, consciousness recovery occurs, and the patient has a certain degree of perception and memory of the surrounding environment or sound. After general anesthesia, the patient can recall what happened during the surgery and be informed of any pain or other conditions. Events occurring before induction to sleep and after awakening from anesthesia were not included.

CONTACTS AND LOCATIONS:
Overall Officials: Min Su, BM, Study Director — First Affiliated Hospital of Chongqing Medical University
Locations (1):
- The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality, China